CLINICAL TRIAL: NCT05999994
Title: CAMPFIRE: Children's and Young Adult Master Protocol for Innovative Pediatric Research
Brief Title: A Master Protocol (LY900023) That Includes Several Clinical Trials of Drugs for Children and Young Adults With Cancer
Acronym: CAMPFIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17304; J1S-MC-JAAA (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms; Child; Adolescent
MeSH Terms: conditions — Neoplasms | interventions — Ramucirumab; Cyclophosphamide; Vinorelbine; Gemcitabine; Docetaxel; abemaciclib; Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Ramucirumab + Cyclophosphamide + Vinorelbine (DSRCT ISA) (Experimental): Ramucirumab given intravenously (IV), cyclophosphamide given orally and vinorelbine given IV in 28-day cycles for desmoplastic small round cell tumor (DSRCT) intervention-specific appendix (ISA).
  Interventions: Drug: Ramucirumab; Drug: Cyclophosphamide; Drug: Vinorelbine
- Cyclophosphamide + Vinorelbine (DSRCT ISA) (Active Comparator): Cyclophosphamide given orally and vinorelbine given IV in 28-day cycles for DSRCT ISA.
  Interventions: Drug: Cyclophosphamide; Drug: Vinorelbine
- Ramucirumab + Gemcitabine + Docetaxel (SS ISA) (Experimental): Ramucirumab and gemcitabine given IV in 21-day cycles for synovial sarcoma (SS) ISA.
  Interventions: Drug: Ramucirumab; Drug: Gemcitabine; Drug: Docetaxel
- Gemcitabine + Docetaxel (SS ISA) (Active Comparator): Gemcitabine and docetaxel given IV in 21-day cycles for SS ISA.
  Interventions: Drug: Gemcitabine; Drug: Docetaxel
- Abemaciclib + Irinotecan + Temozolomide (ES ISA) (Experimental): Abemaciclib given orally, irinotecan given IV, and temozolomide given orally in 21-day cycles for Ewing's sarcoma (ES) ISA.
  Interventions: Drug: Abemaciclib; Drug: Irinotecan; Drug: Temozolomide
- Irinotecan + Temozolomide (ES ISA) (Active Comparator): Irinotecan given IV and temozolomide given orally in 21-day cycles for ES ISA.
  Interventions: Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806
  Arms: Ramucirumab + Cyclophosphamide + Vinorelbine (DSRCT ISA); Ramucirumab + Gemcitabine + Docetaxel (SS ISA)
Drug: Cyclophosphamide — Administered orally
  Arms: Cyclophosphamide + Vinorelbine (DSRCT ISA); Ramucirumab + Cyclophosphamide + Vinorelbine (DSRCT ISA)
Drug: Vinorelbine — Administered IV
  Arms: Cyclophosphamide + Vinorelbine (DSRCT ISA); Ramucirumab + Cyclophosphamide + Vinorelbine (DSRCT ISA)
Drug: Gemcitabine — Administered IV
  Other Names: LY188011
  Arms: Gemcitabine + Docetaxel (SS ISA); Ramucirumab + Gemcitabine + Docetaxel (SS ISA)
Drug: Docetaxel — Administered IV
  Arms: Gemcitabine + Docetaxel (SS ISA); Ramucirumab + Gemcitabine + Docetaxel (SS ISA)
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Abemaciclib + Irinotecan + Temozolomide (ES ISA)
Drug: Irinotecan — Administered IV
  Arms: Abemaciclib + Irinotecan + Temozolomide (ES ISA); Irinotecan + Temozolomide (ES ISA)
Drug: Temozolomide — Administered orally
  Arms: Abemaciclib + Irinotecan + Temozolomide (ES ISA); Irinotecan + Temozolomide (ES ISA)

SUMMARY:
The main purpose of the master is to help the research sites and sponsor carry out several clinical trials more efficiently by providing a common research protocol. Individual clinical trials under this master protocol define drug/disease-specific research goals and activities to test them. New studies will be added as new drugs emerge against different cancers. Participation in the trial will depend on how long the benefit lasts.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the inclusion criteria below. Additional criteria are specified in the protocol amendment (individual addenda) to which the participant will enroll.

* Have either measurable or evaluable disease using standard techniques by the Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).
* The participant has a Lansky (<16 years of age) or Karnofsky (≥16 years of age) performance score of at least 50.
* Participants must have discontinued all previous treatments for cancer or investigational agents greater than or equal to (≥)7 days after the last dose and must have recovered from clinically significant side effects.
* The participant has adequate hematologic and organ function.
* Female participants of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to first dose.
* Both female and male participants of childbearing potential must agree to use highly effective contraceptive precautions during the trial and for at least 3 months following the last dose of study drug.

Participants will be ineligible if they meet any of the exclusion criteria below. Additional criteria are specified in the protocol amendment to which the participant will enroll.

* Participants with severe and/or uncontrolled concurrent medical disease or psychiatric illness/social situation that, in the opinion of the investigator, could cause unacceptable safety risks or compromise compliance with the protocol.
* Participants who have active infections requiring therapy.
* Participants who have had allogeneic bone marrow or solid organ transplant.
* Participants who have had, or are planning to have, certain invasive procedures.
* Female participants who are pregnant or breastfeeding.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-01-22 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Allocated to Each ISA | Baseline up to Week 4
  Number of Participants Allocated to Each ISA

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (66):
- United States (29):
  - Childrens Hospital of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital of Colorado, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Inc. at Egleston, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Washington University Medical School, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Nationwide Children's Hosp, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Cook Children's Hospital, Fort Worth, Texas
  - Texas Childrens Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown
  - Peter MacCallum Cancer Centre, Melbourne
  - Royal Children's Hospital, Melbourne
  - The Sydney Children's Hospitals Network, Westmead
- Belgium (2):
  - UCL- Saint Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- France (3):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Curie, Paris
- Germany (3):
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- Italy (7):
  - IRCCS Istituto Ortopedico Rizzoli, Bologna
  - Istituto di Candiolo IRCCS - Fondazione del Piemonte per l'Oncologia, Candiolo
  - Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Di Padova, Padua
  - Ospedale Bambino Gesu, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (3):
  - National Cancer Center Hospital, Chūōku
  - Kyushu University Hospital, Fukuoka
  - Hyogo Prefectural Kobe Children's Hospital, Kobe
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Prinses Maxima Centrum, Utrecht
- Spain (9):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - University College Hospital - London, London
  - Royal Marsden Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

DOCUMENTS (1):
  • Study Protocol (2019-09-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT05999994/Prot_000.pdf